CLINICAL TRIAL: NCT05663437
Title: Effectiveness of Core Stabilization Exercises With and Without Neural Mobilization Technique in Female Patients With Lumbar Radiculopathy Due to Disc Herniation - an RCT Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Faryah Aslam, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-2696
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Lumbar Disc Herniation
Keywords: Lumbar radiculopathy; Disc herniation; Pain intensity; Functional disability; Core stabilization exerices; Neural mobilization technique; Females
MeSH Terms: conditions — Intervertebral Disc Displacement; Radiculopathy; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Core stabilization exercises
  Interventions: Other: Core stabilization exercises
- Experimental group (Experimental): Core stabilization exercises and Neural mobilization technique
  Interventions: Other: Core stabilization exercises + neural mobilization technique

INTERVENTIONS:
Other: Core stabilization exercises — 6 core stabilization exercises including: dead bug, side lying, prone, bird dog, bridging, planks (1x10 reps for 15-30 secs each exercise) 3 alternative days a week, for 4 weeks.
  Arms: Control group
Other: Core stabilization exercises + neural mobilization technique — 6 core stabilization exercises including: dead bug, side lying, prone, bird dog, bridging, planks (1x10 reps for 15-30 secs each exercise) 3 alternative days a week, for 4 weeks.
  Neural mobilization technique (SLR intervention for first 2 weeks and slider intervention for last 2 weeks).
  Arms: Experimental group

SUMMARY:
Lumbar disc herniation (LDH) is the most frequent cause of lumbosacral radiculopathy and account for 39% of chronic low back pain cases. In approximately 95% of cases LDH occurs at L4-L5 and L5-S1 levels. Maintaining functional stability of lumbar spine necessitates strengthening of the core muscles that plays a key role in lumbar strengthening, motor control and core stability. Core stability may play a role in passive disc stability, reducing the pressure on disc, relieving nerve impingement and radiating pain. Neural mobilization technique involves manual mobilization or exercise that promotes movement between and around the neural structures.This study is intended to add to the existing literature regarding patients with lumbar radiculopathy due to disc herniation, and to report the effectiveness of core stabilization exercises with and without neural mobilization technique in respective population in reduction of associated symptoms, pain and functional disability, enhancing the quality of life, and restoring a prior functional status and activity potential.

DETAILED DESCRIPTION:
An RCT will be conducted on female patients with radiculopathy due to posterolateral disc herniation at L4-S1 levels, visiting Physiotherapy OPD at DUHS Ojha campus. A sample of 70 patients was calculated using PASS v11 software (Microsoft, Redmond, WA, USA). For estimating sample size, pain scores of motor control group (3.4 ±0.9) and motor control+ NDS group (2.5 ±0.8) after 8th session was used from a study conducted earlier. Patients who fulfill the inclusion criteria will be included in the study through convenience sampling, and will be equally allocated either in Core stabilization exercises group A (Control group: n=35) or Core stabilization exercises with Neural mobilization technique group B (Experimental group: n=35). Treatment will be provided on alternate days 3 times a week for 4 consecutive weeks. Patients will be assessed for pain and functional disability prior to the treatment, then at the end of 2nd week and 4th week through 11 points NPRS and Modified Oswestry Disability Questionnaire (MODQ). Data will be entered and analyzed through IBM SPSS version 24 with p-value < 0.05 will be considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed and referred females with lumbar disc herniation.
2. Have a confirmed L4-S1 lumbar disc herniation through an MRI.
3. Postero-lateral Disc herniation of stage I & II.
4. Age group of 30-50 years.
5. Low back pain radiating to one leg for more than 3 months.
6. Positive SLR test reproducing symptoms between 40°-70°.

Exclusion Criteria:

1. Spondylolisthesis, spondylitis, and spinal canal stenosis.
2. Red flags: spinal tumors, cuada equina syndrome, spinal fractures, osteoporosis, infection.
3. Severe vascular disease like DVT.
4. Pregnancy and Gynecological problems.
5. Psychological disorders affecting subject's ability to follow instructions.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 30 -50 years of age
Enrollment: 70 (Estimated)
Dates: Start 2022-10-06 (Actual); Primary Completion 2023-10-05 (Estimated); Study Completion 2023-11-05 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Baseline, 2nd week and 4th week (change is being assessed)
  Numeric Pain Rating Scale (11-point NPRS), a commonly used horizontal line scale with two end points to measure pain intensity. 0 indicates no pain at all, while 10 indicates the worst possible pain experienced.
Functional disability | Baseline, 2nd week and 4th week (change is being assessed)
  Modified Oswestry Disability Questionnaire (MODQ), a self-administered 10 items questionnaire. Items are questions about pain intensity related to activities of daily living. Each section has a score of 0- 5, 5 demonstrating the greatest disability. The percentage of disability is reported by adding scores of all items and multiplying it by 2. Higher score represents higher pain intensity and disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No